CLINICAL TRIAL: NCT06072872
Title: Portable Continuous Positive Airways Pressure (CPAP) in Excessive Central Airway Collapse (ECAC) Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Papworth Hospital NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P03038
Record Dates: First submitted 2023-08-24; First posted 2023-10-10 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Excessive Central Airways Collapse; Respiratory Disease; Tracheobronchomalacia; Excessive Dynamic Airway Collapse
MeSH Terms: conditions — Respiration Disorders; Tracheobronchomalacia

STUDY DESIGN:
Intervention Model Description: Prospective interventional, with first period without use of study device, followed with second period using study device
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No Portable CPAP (No Intervention): Patients continue life as normal without portable CPAP
- Use of portable CPAP (Experimental): Patients use portable CPAP during periods of exercise
  Interventions: Device: Use of portable CPAP

INTERVENTIONS:
Device: Use of portable CPAP — Patients use portable CPAP during exercise
  Arms: Use of portable CPAP

SUMMARY:
This study will investigate the role of a portable Continues Positive Airway Pressure device (pCPAP) in management of patients with symptomatic Excessive Central Airway Collapse (ECAC). ECAC is characterised by complete or partial collapse of central airways on exhalation. In some cases, this can cause persistent breathlessness and severely limited exercise capacity. Current treatment options for ECAC are very limited. Standard assistive breathing devices such as CPAP machines are sometimes used to relieve symptoms at night or at rest. This does not address breathlessness during activity which drives accumulation of disability over time.

The main aims of this project are to assess the effect of a portable CPAP (pCPAP) device on exercise capacity and symptoms and evaluate the feasibility of wearing pCPAP at home during routine activities. Lightweight battery-powered portable CPAP devices have been recently developed to facilitate travel to remote areas by people with Obstructive Sleep Apnoea (OSA). Patients with ECAC can wear them during physical activity to prevent airway collapse but their potential benefits have not been evaluated in clinical trials.

For this study, the investigators will recruit 20 patients with ECAC who will attend for two study visits 4-6 weeks apart in a single centre (The Royal Papworth Hospital). The primary outcome measure will be a shuttle walk test performed repeatedly with and without pCPAP in a randomised order. Secondary outcomes will include assessment of activity level, breathlessness, quality of life ,pCPAP usage and its acceptability. The study will evaluate a pragmatic way of CPAP titration and application. Previously acquired diagnostic baseline computed tomography (CT) scans will be analysed with a novel Functional Respiratory Imaging (FRI) tool. This software tool will enable retrospective reflections on the changes occurring within the lungs for patients with ECAC. This may help identify predictive features of potential pCPAP responders and inform future use.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of ECAC based on >50% reduction of the antero-posterior diameter of large airways demonstrated on dynamic CT thorax or bronchoscopy. Only patients with tracheal and/or bilateral large bronchi (main to lobar) involvement will be included.
2. Symptoms of dyspnoea felt to be predominantly caused by ECAC (where ECAC is the only respiratory pathology or dyspnoea is clearly out of proportion to a co-morbid respiratory condition)
3. Medical Research Council (MRC) breathlessness scale of 3 (I stop for breath after walking about 100 yards or after a few minutes on level ground) or more.
4. Age over 18 years
5. Able to give informed consent -

Exclusion Criteria:

* Patients with dynamic collapse of only segmental airways
* Comorbidity which is likely to be an additional limiting factor in exercise tolerance
* Contraindication to CPAP
* Contraindication to incremental shuttle walk testing (ISWT), including; myocardial infarction within the last 3-5 days, unstable angina, uncontrolled arrhythmia, severe symptomatic cardiac or valvular disease, acute pulmonary embolus, uncontrolled asthma, syncope, mental impairment resulting in inability to perform test.
* Resting oxygen saturations <90% on air or need for ambulatory oxygen therapy
* Immobility that would make ISWT unfeasible
* Severe emphysema
* Acute infectious disease
* Acute respiratory illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-07-27 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
Distance achieved in incremental shuttle walk test with and without portable CPAP | After using portable CPAP for four weeks
  Distance achieved in incremental shuttle walk test with and without portable CPAP after using portable CPAP

SECONDARY OUTCOMES:
Degree of dyspnoea pre and post shuttle walk test | During shuttle walk test performed after four weeks of using portable CPAP
  dyspnoea will be measured using the Borg scale

OTHER OUTCOMES:
Activity levels with and without portable CPAP | 30 day
  Activity levels based on pedometer readings
Average daily usage of CPAP | 30 days
  Absolute hours of daily usage
Quality of life score | 4 weeks
  Respiratory-specific quality of life after use of portable CPAP using St George's Respiratory Questionnaire (scores range from 0 to 100, with higher scores indicating more limitations) and Severe Respiratory Insufficiency (SRI) questionnaire (score of 0 to 100 represents the worst to best health-related quality of life)
Feasibility of CPAP self-titration | 4 weeks
  Feasibility and efficacy of CPAP self-titration using Likert scale (range 1-5, higher scores indicate better outcomes), change in CPAP pressure levels and distance walked whilst using portable CPAP
participant perception of using portable CPAP | 4 weeks
  Participant acceptance of using CPAP and its perceived impact on activity level: assessed using a Likert scale ((range 1-5, higher scores indicate better outcomes)
Correlation between severity of ECAC disease and response to portable CPAP | 4 weeks
  Correlation between severity of ECAC disease (as determined by FRI measurements in CT scans) and response to portable CPAP

CONTACTS AND LOCATIONS:
Overall Officials: Dariusz Wozniak, MD, PhD, Principal Investigator — Royal Papworth Hospital NHS Foundation Trust
Locations (1):
- Royal Papworth Hospital, Cambridge, Cambridgeshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No